CLINICAL TRIAL: NCT04345237
Title: Randomized Clinical Trial on Changes in Body Composition When Ingesting a Dairy Compound Enriched With Leucine Daily for 3 Months
Brief Title: Changes in Body Composition When Ingesting a Dairy Compound Enriched With Leucine
Acronym: LEUCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCAMCFE-00013
Record Dates: First submitted 2020-04-08; First posted 2020-04-14 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-04

CONDITIONS: Elderly Person; Body Composition; Physical Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental group 1 (TS + placebo) (Experimental): Training twice a week, with wave periodization. Traditional training (TS) in two circuits. Each exercise is separated by a rest period of 3 minutes and 5 minutes between circuits.
  Daily consumption for 3 months of placebo milk.
  Interventions: Dietary Supplement: dietary supplement consumption
- Experimental group 2 (TS + leucine) (Experimental): Training twice a week, with wave periodization. Traditional training (TS) in two circuits. Each exercise is separated by a rest period of 3 minutes and 5 minutes between circuits.
  Daily consumption for 3 months of milk enriched with leucine.
  Interventions: Dietary Supplement: dietary supplement consumption
- Experimental group 3 (HRC + placebo) (Experimental): Training twice a week, with wave periodization. High intensity training (HRC) on two circuits. Each exercise is separated by a rest period of 35 seconds and 5 minutes between circuits.
  Daily consumption for 3 months of placebo milk.
  Interventions: Dietary Supplement: dietary supplement consumption
- Experimental group 4 (HRC + leucine) (Experimental): Training twice a week, with wave periodization. High intensity training (HRC) on two circuits. Each exercise is separated by a rest period of 35 seconds and 5 minutes between circuits.
  Daily consumption for 3 months of milk enriched with leucine.
  Interventions: Dietary Supplement: dietary supplement consumption
- Experimental group 5 (no physical exercise + leucine) (Experimental): The subjects will not carry out any type of physical activity.
  Daily consumption for 3 months of milk enriched with leucine.
  Interventions: Dietary Supplement: dietary supplement consumption
- Control (no physical exercise + placebo) (No Intervention): The subjects will not carry out any type of physical activity.
  Daily consumption for 3 months of placebo milk.

INTERVENTIONS:
Dietary Supplement: dietary supplement consumption — Consumption of the product under study for 3 months, milk placebo or experimental product (leucine milk).
  In addition, 5 of the arms perform physical activity training
  Arms: Experimental group 1 (TS + placebo); Experimental group 2 (TS + leucine); Experimental group 3 (HRC + placebo); Experimental group 4 (HRC + leucine); Experimental group 5 (no physical exercise + leucine)

SUMMARY:
Controlled clinical trial, randomized by strata (sex and period of the study), with 6 parallel branches to the study depending on the type of product consumed and the type of physical exercise program performed, double-blind masked for the consumption of the product and single-center.

DETAILED DESCRIPTION:
The subjects that meet the selection criteria will make a total of seven visits to the research laboratory (two of them to collect product) and will carry out the pre-established tests in the protocol. Subsequently, a statistical analysis will be carried out with the variables measured in the study to obtain results.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes with age between 55-70 years.
* Body mass index less than 35.
* Subjects who have given written informed consent to participate in the study.

Exclusion Criteria:

* Consumption during the 6 months prior to the study of functional food enriched with leucine or nutritional supplement based on protein concentrate or that presents in its chemical composition leucine.
* Presence of absolute or relative contraindications ruled by the American College of Sports Medicine (ACSM, 1995), during the performance of stress tests.
* Presence of chronic diseases that prevent the performance of a physical exercise program or an exercise test (disabling arthropathies, moderate / severe chronic lung diseases, ischemic heart disease under treatment, arrhythmias, etc).
* Abuse in the ingestion of alcohol.
* Present hypersensitivity or intolerance to any of the components of the products under study.
* Inability to understand informed consent.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-02-15 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Muscle mass | Change of this measurement at 3 months.
  Dual X-ray absorptiometry (DEXA)
Total fat mass | Change of this measurement at 3 months.
  Dual X-ray absorptiometry (DEXA)
Total fat free mass | Change of this measurement at 3 months.
  Dual X-ray absorptiometry (DEXA)
Fat free mass on upper limb | Change of this measurement at 3 months.
  Dual X-ray absorptiometry (DEXA)
Upper limb fat mass | Change of this measurement at 3 months.
  Dual X-ray absorptiometry (DEXA)
Fat-free mass in the lower limb | Change of this measurement at 3 months.
  Dual X-ray absorptiometry (DEXA)
Lower limb fat mass | Change of this measurement at 3 months.
  Dual X-ray absorptiometry (DEXA)

SECONDARY OUTCOMES:
Elbow extension | This measurement is carried out in each of the groups, at the beginning (baseline) and at 3 months (end).
  Upper limb isokinetic dynamometry. The angular velocities used were 60 ° · s-1 and 270 ° · s-1. The variables measured for each of them were maximum isokinetic torque, maximum isokinetic torque in relation to body weight, total work and average power.
Elbow flexion | This measurement is carried out in each of the groups, at the beginning (baseline) and at 3 months (end).
  Upper limb isokinetic dynamometry. The angular velocities used were 60 ° · s-1 and 270 ° · s-1. The variables measured for each of them were maximum isokinetic torque, maximum isokinetic torque in relation to body weight, total work and average power.
Knee extension | This measurement is carried out in each of the groups, at the beginning (baseline) and at 3 months (end).
  Lower limb isokinetic dynamometry. The angular velocities used were 60 ° · s-1 and 270 ° · s-1. The variables measured for each of them were maximum isokinetic torque, maximum isokinetic torque in relation to body weight, total work and average power.
Knee flexion | This measurement is carried out in each of the groups, at the beginning (baseline) and at 3 months (end).
  Lower limb isokinetic dynamometry. The angular velocities used were 60 ° · s-1 and 270 ° · s-1. The variables measured for each of them were maximum isokinetic torque, maximum isokinetic torque in relation to body weight, total work and average power.
Blood samples: Glycid metabolism and lipid metabolism. | Blood samples will be taken twice, once at baseline, at the beginning of the trial and once at the end after 3 months.
  Basic glucemia, total cholesterol, cholesterol HDL, cholesterol LDL, , triglycerides.
Liver safety variables | Blood samples will be taken twice, once at baseline, at the beginning of the trial and once at the end after 3 months.
  It is a blood test that measures the presence of some enzymes, proteins and bilirubin in the blood, with the aim of determining if there is any alteration in the liver.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain